CLINICAL TRIAL: NCT03318146
Title: Safety, Tolerability and Preliminary Efficacy of Unilateral Latanoprost-loaded Punctual Plug in Patients With Open Angle Early Visual Field Defects Glaucoma or Ocular Hypertension in Comparison to Xalatan © Eye Drops in the Second Eye
Brief Title: Safety, Tolerability and Preliminary Efficacy of Unilateral Latanoprost-loaded Punctual Plug -EXP-LP
Acronym: EXP-LP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXP-LP-1
Record Dates: First submitted 2017-10-02; First posted 2017-10-23 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-09

CONDITIONS: Glaucoma; Ocular Hypertension; IOP
Keywords: Plugged Tear Duct
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Lacrimal Duct Obstruction | interventions — Drug Delivery Systems; Latanoprost

STUDY DESIGN:
Intervention Model Description: The study is a prospective, open-label, controlled non-randomized study, comparative "split body"-design study comparing unilateral Latanoprost-loaded punctual plug in patients with open angle early visual field defects glaucoma or ocular hypertension with Xalatan © eye drops treatment in the second eye.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXP-LP punctum plug (Experimental): EXP-LP is a novel and innovative drug delivery system aiming to improve patient compliance and outcomes. EXP-LP punctum plug, is a non-invasive insert that replaces eye drops and provides sustained therapy for glaucoma, dry eye and other major eye diseases. EXP-LP is a combination of an ophthalmic prostaglandin drug (Latanoprost). The prostaglandin drug works by increasing the natural outflow of fluid from inside the eye
  Interventions: Device: drug delivery system
- XALATAN® (Active Comparator): XALATAN® (latanoprost ophthalmic solution) is an eye drop used to treat high eye pressure/intraocular pressure in people with open-angle glaucoma or ocular hypertension. XALATAN is administrated once a day
  Interventions: Drug: XALATAN®

INTERVENTIONS:
Device: drug delivery system — The EXP-LP sustained released formula inserted into a small punctual plug. The plug is designed to release the drug over a period of up to 6 months in a slow release profile.
  Other Names: punctum plug
  Arms: EXP-LP punctum plug
Drug: XALATAN® — one drop in the affected eye(s) once daily in the evening
  Other Names: latanoprost ophthalmic solution
  Arms: XALATAN®

SUMMARY:
Glaucoma is the most frequent cause of irreversible & preventable blindness worldwide, affecting about 2% of the world's population in people over 40. The major risk factor, and only treatable factor in glaucoma, is increased intraocular pressure (IOP). IOP reduction can slow or arrest the progression of vision loss.

Current treatment consists of drops administered on a daily basis with unfortunately low patient compliance, increasing the chance of blindness.

Eximore's product aims to eliminate the need to apply eye drops on a daily basis and thus solves the significant problem of patient compliance.

DETAILED DESCRIPTION:
Device Description - A combination of punctual plug (new product) as delivery system for Latanoprost (already approved drug). The plug has 2 different sizes of "big plug" (450 µg API) and "small plug" (250 µg API) (Neck diameter of 1.08 mm and 1.06 mm, accordingly) EXP-LP punctum plug is intended to be used as drug delivery system to improve patient compliance and outcomes. EXP-LP is a combination therapy non-invasive insert that replaces eye drops and provides sustained drug therapy for chronic eye problems such as glaucoma.

Xalatan (latanoprost) has been marketed for nearly 15 years, and its performance in reducing IOP is well established Study Design - This is a prospective, single center, open-label, controlled ("split body" design) non-randomized study performed in early visual field defects open angle glaucoma or ocular hypertension patients.

Study Population and Justification - 40 patients with open angle early visual field defects glaucoma (treated with eye drop medications) or ocular hypertension will be enrolled to the study. Due to early feasibility stage of the study, no formal sample size calculation was done for this study.

The intent to treat (ITT) population, defined as enrolled participants including those who leave the study prematurely during the screening period (before EXP-LP insertion).

Handling of Participant Withdrawals - Participants who leave the study prematurely during the screening period (before EXP-LP insertion) will not be replaced and will not be accounted for in the ITT study population. The discontinuing patient will be followed for safety by a phone call, one month after exiting the study. Each case of premature withdrawal will be properly recorded in the Screening Failure Log.

Patient Screening - Prior to any study-related procedure, delegated study team members will approach potentially eligible adult subjects diagnosed with early visual field defects open angle glaucoma or ocular hypertension. Those who may be eligible will be offered the choice of undergoing screening to be enrolled in the study or receiving standard public treatment for their current illness without participating in the study. Subjects who do not meet inclusion criteria or who are for any other reason determined to be too ill for inclusion in the study, or who decline to participate in the study, will be considered and recorded as "screen failure" and receive standard and appropriate treatment.

Informed Consent: The informed consent document will be signed and dated for screening and enrollment and each patient consenting will be documented in the patient medical binder. The patient will be given a copy of the consent form together with the study doctor's letter at the time of enrollment. The clinician will ask the patient about his plans and his willingness to attend all scheduled follow-up visits.

Each patient is considered as a Block unit and each of his eyes is considered the investigational unit. Patients will be identified by a serial number and will be numbered according to their serial recruitment (2 digits).

TRIAL PROCEDURES: All study visits will be performed at morning time (8 a.m. to 10 a.m.) in order to unify measurements and reduce intra-patient variations (across measurements). After informed consent is obtained, a case record form (CRF) including all aspects listed below will be recorded. Eligible patients will be enrolled into the study and will be monitored according to ophthalmic standard examinations.

Visit 1: Screening and pre-insertion washout, as part of pre-operative visit (2-4 weeks before grafting procedure - visit 2)

Following signing of informed consent, potential patients that their treated IOP is lower than 26 mmHg on at least 2 consecutive examinations will be screened for study enrolment by assessment of inclusion and exclusion criteria. The following assessments will be performed:

* Demographics
* Medical history
* Vital signs
* Current medications.
* Sitting IOP (see details below) Eligible patients will be required to stop taking (wash-out) their glaucoma eye-drops medications in both eyes until their IOP level is increased by at least 3 mmHg from start of washout in both eyes Visit 2: Screening & EXP-LP plug insertion in one eye and Xalatan © eye-drops in the second eye, (2 weeks or 4 weeks after beginning washout, visit 2a or 2b accordingly) The below mentioned 3 mmHg increase (inclusion criteria #4) is examined at visit 2a (two weeks after first screening visit) for safety reasons, to ensure the patient "untreated IOP" will be monitored (<31 mmHg for glaucoma patients or < 33 mmHg for ocular hypertension patients).

In case their IOP level is yet to be influenced by the washout (less than 3 mmHG increase), an additional visit (2b, 4 weeks after first screening visit) will be scheduled and performed with the patient. In case the patient IOP was increased by less than 3 mmHG in visit 2b, or either the patient IOP is >30 mmHg for glaucoma patients or >32 mmHg for ocular hypertension patients (exit criteria) that patient will discontinue the study and will be recorded as screening failure.

Once inclusion criteria #4 is verified (either 2a or 2b) study eligibility will be confirmed and the following assessments will be evaluated:

* Vital signs
* Current medications. EXP-LP insertion - As detailed in the Investigator Brochure there will be 2 sizes of the EXP-LP medicated punctual plug: "big" and "small", stored and packed separately. The most suitable size will be pre-defined by the investigator performing the procedure and will be documented in the CRF. The patient will be offered to choose which of his eyes should have the PLUG inserted - limiting investigator bias. The selected eye will be documented in the CRF.

Prior to plug insertion prophylactic topical antibiotic (one eye-drop) will be given to the selected eye.

The plug will be inserted to the lower lacrimal punctum (tear duct) using routine curved eye forceps and under topical anesthesia with drops and using the physician biomicroscope.

Xalatan © administration - the second eye will receive mono-treatment of Xalatan © (Pfizer, latanoprost mono-treatment eye drops) as an internal control. According to the manufacturer's instructions for use - the recommended dosage is one drop once daily. Study administration will be in the evening time. Reduction of the IOP starts approximately 3 to 4 hours after administration and the maximum effect is reached after 8 to 12 hours. Xalatan will be administered by the patient until end of the study, and mis-compliance will be documented in the CRF.

• Study Patient Discharge form - Study qualified personnel will instruct the patient before discharge with specific home instructions and emergency contact numbers.

Short-term follow up visits:

Visit 3-8: clinical and biomicroscope examinations (see appropriate time windows below)

The following assessments will be performed during each visit at the hospital clinic:

* Vital signs
* Current medications.
* Sitting IOP The patient will be asked to report any ophthalmic complication: for example: Intraocular inflammation, ocular redness, eyelid edema and hyperaemia conjunctival erythema (see anticipated complications list above) - all will be investigated by the sub-investigator using Visit safety Follow-Up Form. In addition, the patient will be questioned regarding his general morbidity, any other Adverse Events and concomitant medications.

Plug tolerability follow-up - During each visit, placement of plug will be verified. If the plug is not visualized or if the subject is inconvenienced by the inserted plug, the investigator can choose to insert another plug with a different size up to a maximum of 3 replacements.

1. The plug should not be reinserted in case a moderate to serious AE is observed, e.g. rejection or immune reaction, moderate to severe conjunctival hyperemia, moderate to severe Intraocular inflammation, corneal Keratitis (see Table 5, State of the Art Safety Risks, Latanoprost for Glaucoma, Literature Based; Causes, Mitigation & Relation to EXP-LP plug).
2. Any of the following AEs: initial irritation, local discomfort, increased lacrimation, dry eye, mild conjunctival hyperemia, mild Intraocular inflammation or blepharitis may be resolved within a week - treatment with lubricating drops or topical antibiotics maybe consider according to the physician judgment. In case of persistent occurrence the plug will be replaced with a smaller type if applicable Each replacement will be reported in the CRF.

Visit 8: Investigational EXP-LP plug removal (termination): (3 months (+\- 7 days) from plug insertion) In addition to the above mentioned study evaluations, EXP-LP plug will be removed by study qualified investigator under prior topical prophylactic antibiotic (one eye-drop) topical anaesthesia drops, using a biomicroscope and routine curved eye forceps. Intactness of the plug will be examined and recorded in the CRF

• Study Termination form - Study qualified personnel will instruct the patient before discharge with specific medication instructions and prescriptions for both eyes.

Un-scheduled visit:

The study investigator will instruct the patient to immediately contact the study team in case of: plug loss, intraocular inflammation, eyelid edema and keratitis.

The patient must call the study nurse to schedule an un-scheduled visit which may only be performed by one of the study investigators, and will be reported to the principal investigator.

For unscheduled visits the patient will be clinically managed by the study team with additional full eyes examination to be done at the discretion of the investigator.

Data Monitoring and Quality Control - The investigator, through an appointed Clinical Research Associate (CRA), will be responsible for implementing and maintaining quality assurance and quality control systems with written Standard Of Procedures to ensure that trials are conducted and data are generated, documented (recorded), and reported in compliance with the protocol, GCP, and the applicable regulatory requirement(s), including ISO 14155:2011.The investigator will be responsible for ensuring direct access to all trial related sites, source data/documents, and reports for the purpose of monitoring and auditing by the hospital, and inspection by Israeli regulatory authorities. Quality control should be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly. The study CRA will verify that (a) The rights and well-being of human patients are protected, (b) The reported trial data are accurate, complete, and verifiable from source documents and (c) The conduct of the trial is in compliance with the currently approved protocol/amendment(s), with GCP, and with the applicable regulatory requirement(s) (including ISO 14155:2001). The monitor will submit a written report after each trial-site visit or trial related communication. A report should include the date, site, name of the monitor, and name of the investigator or other individual(s) contacted. A report should include a summary of what the monitor reviewed and the monitor's statements concerning the significant findings/facts, deviations and deficiencies, conclusions, actions taken or to be taken and/or actions recommended to secure compliance. To ensure compliance of this investigator initiated trial with current national regulations and the ICH guidelines, data generated by this study will be available for inspection upon request by representatives of the local health authorities- IRB or the national authorities - MOH, or any entity providing support for this trial. The general scope of such visits would be to inspect study data (regulatory requirements), source documentation and CRF completion in accordance with current GCP, the ICH guidelines and the respective local and national government regulations and guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years consecutive males or females diagnosed with open angle early visual field defects glaucoma or ocular hypertension in both eyes and treated with eye drop medications .
2. Treated IOP lower than 26 mmHg on at least 2 consecutive examinations.
3. If glaucoma, mean deviation must be better than -10 mmHg in study eye (early visual field defects glaucoma)
4. IOP increase of at least 3 mmHg from start of washout in both eyes.

   Exclusion Criteria:
5. Any record of IOP ever being higher than 33 mmHg.
6. Corneal or other anatomical abnormalities preventing reliable applanation tonometry
7. Severe dry eye,
8. Use of contact lenses
9. Intolerance or contraindication to latanoprost or BAK
10. Indication of optic nerve damage and visual function deterioration according to the investigator's judgment
11. Lower lacrimal Punctum (tear duct) diameter is smaller than 0.4mm or greater than or equal to 0.75mm
12. Pregnancy or lactation (questioned by the consenting investigator), unwillingness to avoid pregnancy
13. Use of (topical or systemic) corticosteroids within 2 months before enrolment. Any systemic condition or medication that can affect IOP.
14. Known intolerance to PGA eye drops
15. Use of oral IOP-lowering medication
16. Punctual occlusions or other anatomic abnormality
17. Previous incisional ocular surgery (e.g., conventional filtering surgery) to lower IOP
18. Evidence of current or prior angle closure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint - the incidence of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v4.0. | Will be evaluated through study completion (3 months)
  Main Adverse Event that will be focused on during the study:
  * Irritation and local discomfort
  * Increased Lacrimation
  * Increased mucus
  * Intraocular inflammation
  * Ocular redness
  * Eyelid Edema
  * Hyperaemia conjunctival erythema
  * Keratitis

SECONDARY OUTCOMES:
Tolerability Endpoint - The incidence of subjects withdrew due to plug inconvenience and plug incompatibility | Will be evaluated through study completion (3 months)
  Tolerability will be evaluated on the basis of withdrawal rates over time.

OTHER OUTCOMES:
Exploratory Endpoint - (preliminary efficacy): To demonstrate the performance in lowering IOP of EXP-LP in comparison to Xalatan © eye drops treatment in the second eye. | Will be evaluated through study completion (3 months)
  Endpoints will be IOP differences from baseline of:
  i. The plug inserted eye compared to the controlled treated eye at all study follow-up visits ii. The plug inserted eye at all study follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Tal Lavi, Study Director — Gsap Medical Ltd.; Ishay Attar, CEO, Study Chair — Eximore Ltd.
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No
IPD is not intended to be shared as this will be a single site study. The study will be public at ClinicalTrial.gov

REFERENCES:
- [Result] Boland MV, Ervin AM, Friedman DS, Jampel HD, Hawkins BS, Vollenweider D, Chelladurai Y, Ward D, Suarez-Cuervo C, Robinson KA. Comparative effectiveness of treatments for open-angle glaucoma: a systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2013 Feb 19;158(4):271-9. doi: 10.7326/0003-4819-158-4-201302190-00008. PMID 23420235
- [Result] Burr J, Azuara-Blanco A, Avenell A, Tuulonen A. Medical versus surgical interventions for open angle glaucoma. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD004399. doi: 10.1002/14651858.CD004399.pub3. PMID 22972069
- [Result] Chen R, Yang K, Zheng Z, Ong ML, Wang NL, Zhan SY. Meta-analysis of the Efficacy and Safety of Latanoprost Monotherapy in Patients With Angle-closure Glaucoma. J Glaucoma. 2016 Mar;25(3):e134-44. doi: 10.1097/IJG.0000000000000158. PMID 25383466
- [Result] Cucherat M, Stalmans I, Rouland JF. Relative efficacy and safety of preservative-free latanoprost (T2345) for the treatment of open-angle glaucoma and ocular hypertension: an adjusted Indirect comparison meta-analysis of randomized clinical trials. J Glaucoma. 2014 Jan;23(1):e69-75. doi: 10.1097/IJG.0b013e3182a075e6. PMID 23881267
- [Result] Eveleth D, Starita C, Tressler C. A 4-week, dose-ranging study comparing the efficacy, safety and tolerability of latanoprost 75, 100 and 125 mug/mL to latanoprost 50 mug/mL (xalatan) in the treatment of primary open-angle glaucoma and ocular hypertension. BMC Ophthalmol. 2012 May 18;12:9. doi: 10.1186/1471-2415-12-9. PMID 22607109
- [Result] Garway-Heath DF, Crabb DP, Bunce C, Lascaratos G, Amalfitano F, Anand N, Azuara-Blanco A, Bourne RR, Broadway DC, Cunliffe IA, Diamond JP, Fraser SG, Ho TA, Martin KR, McNaught AI, Negi A, Patel K, Russell RA, Shah A, Spry PG, Suzuki K, White ET, Wormald RP, Xing W, Zeyen TG. Latanoprost for open-angle glaucoma (UKGTS): a randomised, multicentre, placebo-controlled trial. Lancet. 2015 Apr 4;385(9975):1295-304. doi: 10.1016/S0140-6736(14)62111-5. Epub 2014 Dec 19. PMID 25533656
- [Result] Kompella UB, Kadam RS, Lee VH. Recent advances in ophthalmic drug delivery. Ther Deliv. 2010 Sep;1(3):435-56. doi: 10.4155/TDE.10.40. PMID 21399724
- See also: NCI Common Terminology Criteria for Adverse Events — http://evs.nci.nih.gov/ftp1/CTCAE/About.html